CLINICAL TRIAL: NCT03825614
Title: Does The Pilates or Therapeutic Exercises Effects on Functional Level, Depression, Pain, Qualıty of Life in Young Adults
Brief Title: The Effect of Exercises on Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, asuman saltan, ASSIST PROF, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UYalova
Record Dates: First submitted 2019-01-04; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Exercise; Young Adults; Quality of Life; Pain; Depressive Symptoms
MeSH Terms: conditions — Motor Activity; Pain; Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- training gruop (Experimental): The plates exercise program is concerned with the following main principles: efficient breathing, mental concentration, relaxation, correct spine elongation and posture, correct abdominal muscle control over spine stability and mobility, correct function of each upper and lower limb, precision, lowing integrated movement, and achieving muscle strength and stamina.
  Interventions: Behavioral: training
- training group (Active Comparator): Therapeutic exercise program was designed according to the American Collage of Sports Medicine's recommendations for healthy people. The exercise program was conducted using low- to moderate-intensity therapeutic exercises. These therapeutic exercises included a short educational talk that provided information on proper body mechanics, the benefits of exercise, realistic goal-setting, and overcoming common barriers (such as fear) when developing an exercise routine.
  Interventions: Behavioral: training
- Control group (No Intervention): Participants in the control group have no exercise in this study.

INTERVENTIONS:
Behavioral: training — plates and therapeutic exercises applied on young adults
  Arms: training group; training gruop

SUMMARY:
The aim of this study was to assess the treatment effect of plates and conventional exercises on health related quality of life, pain, functional level, psychological state in young adults. Randomised controlled study. Participants were randomly divided into 3 groups: a plates exercise group (n = 29), a therapeutic exercise group (n = 21), and a control group (n = 35). The therapeutic and plates groups underwent related training programs for 3 month, while the controls had no specific training. After demographic knowledge were collected the investigators carried out the following assessments on all participants: the Visual Analog Scale (VAS), Waist/ Hip ratio (WHr), Beck Depression Inventory (BDI), Oswestry Disability Index (ODI), Notthingham Health Profile (NHP). All subjects were evaluated at baseline and post-training.

ELIGIBILITY:
Inclusion Criteria:

• They were apparently healthy and had no systematic diseases or any problem preventing their participation in any exercise program.

Exclusion Criteria:

* Having a systemic pathology, including inflammatory, rheumatologic, or metabolic diseases
* Having any musculoskeletal injury, pathology, or structural deformity related to the spine or extremities
* Having any active intervention including corticosteroid or any medication in the previous 3 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in the pain | 12 weeks
  A visual analogue scale (VAS) was used to their level of pain subjects experienced throughout these activities. The VAS is comprised of a 10 cm horizontal line, wherein 0 indicates "no pain" and 10 indicates "unbearable pain" (Sang, Sang, Dong and Byung, 2016). Participants were asked to mark the strength of their ongoing musculoskeletal pain on the horizontal line.
Assessment of changes in the depression | 12 weeks
  The Back Depression Inventory (BDI) was used to determine patients' level of depression; each item on the scale is given a score of one to three, allowing for a maximum test score of 63 according to form. A subjects' total overall score is then used as an indicator of the presence and severity of depression: a total score lower than 10 indicates no depression, a score of 10-17 indicates mild depression, a score of 18-29 indicates moderate-to-severe depression, and a score of 30 or above indicates severe depression (Muyan, Sancak and Demir, 2017).
Health related quality of life | 12 weeks
  The Turkish version of the Nottingham Health Profile (NHP) was used to assess participants' health-related quality of life. The NHP is a general quality of life questionnaire that measures individuals' perceived health problems and the extent to which these problems affect their normal daily activities. The questionnaire is comprised of 38 items and evaluates six dimensions of healthy individuals' health statuses, these include: energy (three items), pain (eight items), emotional reactions (nine items), sleep (five items), social isolation (five items) and physical activity (eight items). The test includes a list of yes/no questions. Each section yields a score between 0 and 100 for each subject, where 0 represents the best possible health status and 100 represent the worst possible health status (Liang, Wang and Tao, 2015).
Functional level | 12 weeks
  The Oswestry Disability Index (ODI) questionnaires were distributed to participants and scored according to the study by Yakut et al. The research authors noted that some of the questions on the ODI are directly related to physical activities (lifting, walking, etc.). The level of disability was evaluated using the ODI, which is a condition specific questionnaire regarding how low back pain affects activities of daily living. The questionnaire rates 10 different activities based on a six-point scale, with 0 for ''no pain at all'' and 5 for ''cannot perform due to pain''. The higher the score, the greater the disability the subject was deemed to have (Rodríguez-Romero, Bello, Vivas Costa and Carballo-Costa, 2018).
Assessment of changes in the Waist and Hip circumference | 12weeks
  To find the waist/hip (WHr) ratio, participants' waist circumference was taken in centimeters (cm) using a tape measure to measure the point midway between the costal margin and iliac crest on the mid-axillary line, with the subject standing and breathing normally. Hip circumference (cm) was measured at the widest point around the greater trochanter. The waist-to-hip ratios of participants were calculated by dividing their waist measurement by their hip measurement (Tam and Çakır, 2012).

CONTACTS AND LOCATIONS:
Overall Officials: saltan, Principal Investigator — researcher

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toprak Celenay S, Ozer Kaya D. An 8-week thoracic spine stabilization exercise program improves postural back pain, spine alignment, postural sway, and core endurance in university students:a randomized controlled study. Turk J Med Sci. 2017 Apr 18;47(2):504-513. doi: 10.3906/sag-1511-155. PMID 28425239
- [Result] Caldwell K, Harrison M, Adams M, Triplett NT. Effect of Pilates and taiji quan training on self-efficacy, sleep quality, mood, and physical performance of college students. J Bodyw Mov Ther. 2009 Apr;13(2):155-63. doi: 10.1016/j.jbmt.2007.12.001. Epub 2008 Feb 20. PMID 19329051
- [Result] Ozer Kaya D, Duzgun I, Baltaci G, Karacan S, Colakoglu F. Effects of calisthenics and Pilates exercises on coordination and proprioception in adult women: a randomized controlled trial. J Sport Rehabil. 2012 Aug;21(3):235-43. doi: 10.1123/jsr.21.3.235. Epub 2011 Nov 16. PMID 22104298